CLINICAL TRIAL: NCT01794182
Title: A Randomized, Multi-Center, Prospective, Double Blind, Phase II Trial of RP- 1127 (Glyburide for Injection) in Patients With a Severe Anterior Circulation Ischemic Stroke Who Are Likely to Develop Malignant Edema
Brief Title: Glyburide Advantage in Malignant Edema and Stroke - Remedy Pharmaceuticals
Acronym: GAMES-RP
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Remedy Pharmaceuticals, Inc. (Industry)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Quadruple | Purpose: Prevention
Other Study IDs: 252LH203; RPI 203 (Other: Remedy Pharmaceuticals, Inc.)
Record Dates: First submitted 2013-02-14; First posted 2013-02-18 (Estimated); Last update posted 2024-11-12 (Actual); Status verified 2024-11

CONDITIONS: Ischemic Stroke; Malignant Edema
MeSH Terms: conditions — Ischemic Stroke; Anthrax | interventions — Glyburide; Injections

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator, Outcomes Assessor
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- Matching Placebo (Placebo Comparator): Participants received a bolus dose of matching placebo over 2 minutes, followed by a continuous matching placebo infusion for 72 hours.
  Interventions: Drug: Placebo
- Glyburide for Injection (Experimental): Participants received a 0.13 mg bolus dose of glyburide over 2 minutes, followed by a 0.16 mg/hr continuous infusion for 6 hours and than a 0.11 mg/hr for 66 hours for a total dosing period of 72 hours.
  Interventions: Drug: Glyburide for Injection

INTERVENTIONS:
Drug: Glyburide for Injection — Administered as specified in the treatment arm.
  Other Names: RP-1127; glibenclamide; glybenclamide
  Arms: Glyburide for Injection
Drug: Placebo — Administered as specified in the treatment arm.
  Arms: Matching Placebo

SUMMARY:
This is a randomized, multi-center, prospective, double blind study. The primary objective is to assess the efficacy and safety of glyburide (RP-1127) compared to placebo in participants with a severe anterior circulation ischemic stroke who are likely to develop malignant edema.This objective will be addressed by comparing the proportion of glyburide treated particpants and placebo treated participants with a Day 90 modified Rankin Scale (mRS) ≤ 4 without decompressive craniectomy (DC). The secondary objective is to assess the efficacy of RP-1127 compared to placebo in participants with a severe anterior circulation ischemic stroke who were likely to develop malignant edema.

DETAILED DESCRIPTION:
The study population consists of participants with a clinical diagnosis of acute severe anterior circulation ischemic stroke, a baseline diffusion weighted image (DWI) lesion between 82 and 300 cm3, age 18-80 years, and time from symptom onset to start of study infusion of ≤10 hours. The study will enroll both participants that do not receive intravenous (IV) recombinant tissue plasminogen activator (rtPA) and those that receive IV rtPA within 4.5 hours of stroke.

Enrollment will be randomized controlling for site, age ≤60 (yes/no), and IV rtPA treatment at baseline (yes/no). Participants will be randomized equally between glyburide and placebo.

ELIGIBILITY:
Key Inclusion Criteria:

* A clinical diagnosis of acute ischemic stroke in the MCA territory (PCA and/or ACA territory involvement in addition to primary MCA territory stroke is acceptable).
* Prior to stroke, no disability, or no significant disability despite symptoms (able to carry out all usual duties and activities).
* A baseline DWI lesion between 82 and 300 cm3 on MRI.
* Patients treated with IV rtPA should meet established criteria for IV rtPA administration in the 0-3 and 3-4.5 hr time periods at the time of rtPA administration (if rtPA is administered in the 3-4.5 hr time window, the NIHSS must be ≤ 25 at the time of rtPA administration).
* The time to the start of infusion of Study Drug must be ≤ 10 hours after time of symptom onset, if known, or the time last seen well [termed "time last known at neurologic baseline" (TLK@B)].
* Provision of written informed consent by a legally authorized representative according to institutional guidelines and national regulations.

Key Exclusion Criteria:

* Commitment to decompressive craniectomy (DC) prior to enrollment, or following enrollment and prior to start of Study Drug.
* Treatment with intra-arterial (IA) rtPA or by mechanical means for clot disruption.
* Patients unable to tolerate MRI scanning, e.g. those with pacemakers or automatic defibrillators.
* Evidence (clinical or imaging) of concurrent infarction in the contralateral hemisphere deemed by the investigator to be sufficiently serious so as to affect functional outcome.
* Clinical signs of herniation, e.g. one or two dilated, fixed pupils; unconsciousness (i.e., ≥ 2 on item 1a on the NIHSS); and/or loss of other brain stem reflexes attributable to edema or herniation according to the investigator's judgment.
* Hemorrhage (other than small petechial hemorrhages) on CT/MRI, or CT/MRI evidence of anteroseptal/pineal shift greater ≥2 mm prior to enrollment that is due to cerebral edema.
* Severe renal disorder from the patient's history (e.g. dialysis) or eGFR of < 30 mL/min/1.73 m2.
* Severe liver disease or ALT >3 times normal, or bilirubin >2 times normal.
* Blood glucose <55 mg/dL at enrollment or immediately prior to administration of Study Drug, or a clinically significant history of hypoglycemia.
* Acute ST elevation myocardial infarction, and/or acute decompensated HF, and/or QTc>520 ms, and/or known history of cardiac arrest (PEA, VT, VF, asystole), and/or admission for an ACS, MI, or coronary intervention (PCI or coronary artery surgery) within the past 3 months.
* Known sulfonylurea treatment within 7 days. Sulfonylureas include glyburide /glibenclamide (Diabeta, Glynase); glyburide plus metformin (Glucovance); glimepiride (Amaryl); repaglinide (Prandin); netaglinide (Starlix); glipizide (Glucotrol, GlibeneseR, MinodiabR); gliclazide (DiamicronR); tolbutamide (Orinase, Tolinase); glibornuride (Glutril).
* Known allergy to sulfa or specific allergy to sulfonylurea drugs.
* Known G6PD enzyme deficiency.
* Pregnant women. Women must be either post-menopausal (as confirmed by the LAR), permanently sterilized or, if ≤ 50 years old must have a negative test for pregnancy obtained before enrollment.
* Breast-feeding women who do not agree (or their LAR does not agree) to stop breast- feeding during Study Drug infusion and for 7 days following the end of Study Drug infusion.
* Patients already enrolled in a non-observation-only stroke study, or with life-expectancy <3 months not related to current stroke, or those unlikely to be compliant with follow up.
* Patients currently receiving an investigational drug.
* Patients in whom a peripheral IV line cannot be placed.
* Mentally incompetent (prior to qualifying stroke) patients and wards of the state.
* Patients who, in the opinion of the investigator, are not suitable for the study (reason to be documented).

NOTE: Other protocol defined inclusion/exclusion criteria may apply

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 86 (Actual)
Dates: Start 2013-06-13 (Actual); Primary Completion 2016-04-04 (Actual); Study Completion 2016-04-04 (Actual)

PRIMARY OUTCOMES:
Percentage of Participants with a Modified Rankin Scale (mRS) score of ≤ 4 Without Decompressive Craniectomy (DC) | Day 90
  The mRS scale runs from 0-6, the scoring is as follows: 0 - No symptoms, 1 - No significant disability, 2 - Slight disability, 3 - Moderate disability, 4 - Moderately severe disability, 5 - Severe disability, 6 - Dead
Number of Participants with Adverse Events and Serious Adverse Events | Up to 1 Year
  An adverse event (AE) is any symptom, sign, illness or experience that develops or worsens in severity during the course of the study. A serious adverse event is any AE that is fatal, life-threatening, requires or prolongs hospital stay, results in persistent or significant disability or incapacity, a congenital anomaly or birth defect, or an important medical event

SECONDARY OUTCOMES:
Percentage of Participants Undergoing DC or Dead | Baseline and Day 14
Change from Baseline in Ipsilateral Hemispheric Swelling | Baseline up to 72-96 Hours
  To be assessed using Magnetic Resonance Imaging (MRI).
Change from Baseline in Lesional Swelling | Baseline up to 72-96 Hours
  To be assessed using MRI.

CONTACTS AND LOCATIONS:
Overall Officials: Medical Director, Study Director — Remedy Pharmaceuticals
Locations (17):
- United States (17):
  - University of Arizona Medical Center, Tucson, Arizona
  - Stanford University Medical Center, Stanford, California
  - Yale University School of Medicine, New Haven, Connecticut
  - University of Florida, Jacksonville, Jacksonville, Florida
  - Northwestern Memorial Hospital, Chicago, Illinois
  - University of Louisville Hospital, Louisville, Kentucky
  - Maine Medical Center, Scarborough, Maine
  - University of Maryland School of Medicine, Baltimore, Maryland
  - Massachusetts General Hospital, Boston, Massachusetts
  - UMASS Memorial Medical Center, Worcester, Massachusetts
  - Cleveland Clinic, Cleveland, Ohio
  - Ohio State University Wexner Medical Center, Columbus, Ohio
  - Oregon Health & Science University Hospital, Portland, Oregon
  - Abington Memorial Hospital, Abington, Pennsylvania
  - UPMC Presbyterian Hospital, Pittsburgh, Pennsylvania
  - Medical University of South Carolina, Charleston, South Carolina
  - University of Utah Healthcare, Salt Lake City, Utah

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Payabvash S, Falcone GJ, Sze GK, Jain A, Beslow LA, Petersen NH, Sheth KN, Kimberly WT. Poor Outcomes Related to Anterior Extension of Large Hemispheric Infarction: Topographic Analysis of GAMES-RP Trial MRI Scans. J Stroke Cerebrovasc Dis. 2020 Feb;29(2):104488. doi: 10.1016/j.jstrokecerebrovasdis.2019.104488. Epub 2019 Nov 29. PMID 31787498
- [Derived] Vorasayan P, Bevers MB, Beslow LA, Sze G, Molyneaux BJ, Hinson HE, Simard JM, von Kummer R, Sheth KN, Kimberly WT. Intravenous Glibenclamide Reduces Lesional Water Uptake in Large Hemispheric Infarction. Stroke. 2019 Nov;50(11):3021-3027. doi: 10.1161/STROKEAHA.119.026036. Epub 2019 Sep 20. PMID 31537189
- [Derived] Kimberly WT, Bevers MB, von Kummer R, Demchuk AM, Romero JM, Elm JJ, Hinson HE, Molyneaux BJ, Simard JM, Sheth KN. Effect of IV glyburide on adjudicated edema endpoints in the GAMES-RP Trial. Neurology. 2018 Dec 4;91(23):e2163-e2169. doi: 10.1212/WNL.0000000000006618. Epub 2018 Nov 16. PMID 30446594
- [Derived] Sheth KN, Petersen NH, Cheung K, Elm JJ, Hinson HE, Molyneaux BJ, Beslow LA, Sze GK, Simard JM, Kimberly WT. Long-Term Outcomes in Patients Aged </=70 Years With Intravenous Glyburide From the Phase II GAMES-RP Study of Large Hemispheric Infarction: An Exploratory Analysis. Stroke. 2018 Jun;49(6):1457-1463. doi: 10.1161/STROKEAHA.117.020365. Epub 2018 May 22. PMID 29789393
- [Derived] Sheth KN, Elm JJ, Molyneaux BJ, Hinson H, Beslow LA, Sze GK, Ostwaldt AC, Del Zoppo GJ, Simard JM, Jacobson S, Kimberly WT. Safety and efficacy of intravenous glyburide on brain swelling after large hemispheric infarction (GAMES-RP): a randomised, double-blind, placebo-controlled phase 2 trial. Lancet Neurol. 2016 Oct;15(11):1160-9. doi: 10.1016/S1474-4422(16)30196-X. Epub 2016 Aug 23. PMID 27567243